CLINICAL TRIAL: NCT02401815
Title: A Phase 1b and 2a Study to Assess Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of CGT9486 as a Single Agent and in Combination With PLX3397 or Sunitinib (Sutent®) in Patients With Advanced Solid Tumors and Patients With Locally Advanced, Unresectable, or Metastatic Gastrointestinal Stromal Tumor (GIST) Who Have Been Previously Treated With Imatinib Mesylate/KIT-Directed Tyrosine Kinase Inhibitor (TKI) Therapy
Brief Title: CGT9486 (Formerly Known as PLX9486) as a Single Agent and in Combination With PLX3397 (Pexidartinib) or Sunitinib in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cogent Biosciences, Inc. (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLX121-01
Record Dates: First submitted 2015-03-19; First posted 2015-03-30 (Estimated); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; KIT; Biomarkers; PLX9486; PLX3397; Sunitinib; CGT9486; GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — pexidartinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1: CGT9486 250 mg QD (Experimental): Participants will receive CGT9486 250 milligrams (mg) orally once daily (QD) in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486
- Part 1: CGT9486 350 mg QD (Experimental): Participants will receive CGT9486 350 mg orally QD in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486
- Part 1: CGT9486 500 mg QD (Experimental): Participants will receive CGT9486 500 mg orally QD in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486
- Part 1: CGT9486 1000 mg QD (Experimental): Participants will receive CGT9486 1000 mg orally QD in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486
- Part 1: CGT9486 500 mg BID (Experimental): Participants will receive CGT9486 500 mg orally twice daily (BID) in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486
- Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) (Experimental): Participants in fasting condition will receive CGT9486 500 mg orally QD in combination with pexidartinib 600 mg (administered as 1 capsule of 200 mg in the morning and 2 capsules of 200 mg in the evening) orally in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486; Drug: Pexidartinib
- Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) (Experimental): Participants in non-fasting condition will receive CGT9486 500 mg orally QD in combination with pexidartinib 600 mg (administered as 1 capsule of 200 mg in the morning and 2 capsules of 200 mg in the evening) orally in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486; Drug: Pexidartinib
- Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg (Experimental): Participants will receive CGT9486 500 mg orally QD in combination with sunitinib 25 mg orally in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486; Drug: Sunitinib
- Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg (Experimental): Participants will receive CGT9486 1000 mg orally QD in combination with sunitinib 25 mg orally in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486; Drug: Sunitinib
- Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg (Experimental): Participants will receive CGT9486 1000 mg orally QD in combination with sunitinib 37.5 mg orally in 28-day dosing cycles. Treatment will continue until participant discontinuation, withdrawal, or study termination.
  Interventions: Drug: CGT9486; Drug: Sunitinib

INTERVENTIONS:
Drug: CGT9486 — CGT9486 will be administered per dose and schedule specified in the arm.
Drug: Pexidartinib — Pexidartinib capsules will be administered per dose and schedule specified in the arm.
  Other Names: PLX3397
  Arms: Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting); Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting)
Drug: Sunitinib — Sunitinib will be administered per dose and schedule specified in the arm.
  Arms: Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg; Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg; Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg

SUMMARY:
The goal of this clinical research study is to learn how CGT9486 (fka PLX9486) may affect cancer cells with certain mutations in the KIT gene, specifically in participants with types of advanced solid tumors including gastrointestinal stromal tumor (GIST).

CGT9486 (fka PLX9486) is designed to block KIT gene mutations. These mutations can cause cancer and cancer cell growth. By blocking these mutations, the drug may kill the cancer cells with the mutation and/or stop the tumor from growing. By combining CGT9486 (fka PLX9486) with PLX3397 and CGT9486 (fka PLX9486) with sunitinib, the investigators hope to block most KIT gene mutations that drive cancer growth.

DETAILED DESCRIPTION:
This study includes a dose escalation portion (Part 1) in which the safety profile and recommended phase 2 dose (RP2D) of CGT9486 as a single oral agent will be evaluated in participants with solid tumors (including GIST), followed by signal-seeking extension cohorts (Part 2). Enrollment in the combination treatment portions of the study (dose-finding for the CGT9486 + pexidartinib combination [Part 2b] and the CGT9486 + sunitinib combination [Part 2e]) is planned to be accrued using standard 3+3 study designs.

Parts 2a, 2c, 2d, and 2f are not conducted due to business decisions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old.
* Part 1, Part 2b, Part 2d, and Part 2e: Participants with advanced solid tumors who have tumor progression following standard therapy, have treatment-refractory disease, or for whom there is no effective standard of therapy.
* Part 2d: Participants with non GIST solid tumors with KIT mutations, who are TKI naïve or have been previously treated with KIT directed TKI therapy who are appropriate for KIT directed TKI therapy
* Part 2a, Part 2c, and Part 2f (GIST participants): Histologically confirmed locally advanced, metastatic and/or unresectable GIST.
* Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test at Screening (≤7 days prior to the first dose of study drug) and must agree to use an effective form of contraception from the time of the negative pregnancy test up to 6 months after the last dose of study drug.
* Fertile men must agree to use an effective method of birth control during the study and for up to 6 months after the last dose of study drug.
* All associated toxicity from previous or concurrent cancer therapy must be resolved (to ≤ Grade 1 or Baseline) prior to study treatment administration.
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Life expectancy ≥3 months.
* Adequate hematologic, hepatic, and renal function:
* Left ventricular ejection fraction (LVEF) >50% per echocardiogram (ECHO) or multiple-gated acquisition (MUGA) for participants on the sunitinib arms (Parts 2e and f).

Exclusion Criteria:

* Known or demonstrated wild type KIT or platelet-derived growth factor receptors (PDGF-R), or known or demonstrated mutations of PDGF R, sorbitol dehydrogenase (SDH), or neurofibromin 1 (NF 1) that are causative for the observed malignancy.
* For Part 1 (phase 1, single agent): Participants with a known or presumed pathogenic KIT exon 13 or 14 resistance mutation.
* Parts 2a and 2d: Participants with known or presumed pathogenic KIT exon 13 or 14 resistance mutations. (However, such participants are permitted on the combination arms of Parts 2b, 2c, 2e, or 2f.)
* Presence of symptomatic or uncontrolled brain or central nervous system metastases. Participants with stable, treated brain metastases are eligible for this trial. However, participants must not have required steroid treatment for their brain metastases within 30 days of Screening.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.
* Clinically significant cardiac disease
* Inability to take oral medication or significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption.
* Ongoing infection of ≥ Grade 2 severity.
* Non-healing wound, ulcer, or bone fracture.
* Known human immunodeficiency virus (HIV)-positive individuals on combination antiretroviral therapy, participants with known active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy
* Hepatobiliary diseases including biliary tract diseases, autoimmune hepatitis, inflammation, fibrosis, or cirrhosis of liver caused by viral, alcohol, or genetic reasons. Gilbert's disease is allowed if total bilirubin is ≤1.5 * upper limit of normal (ULN).
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Females who are pregnant or nursing.
* Any psychological, familial, sociological, or geographical condition that could hamper compliance with the study protocol.
* Strong CYP3A4 inhibitors or inducers within 14 days or 5 drug half-lives of the agent, whichever is longer, of study drug initiation or the need to continue these drugs during this study.
* Major surgery or significant traumatic injury within 14 days of Cycle 1 Day 1.
* History (within 2 years prior to first study drug administration) of another malignancy unless the malignancy was treated with curative intent and likelihood of relapse is small (<5% in 2 years in the judgment of the investigator).
* Anti-cancer therapy within the period immediately before Cycle 1 Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sachs, MD, Study Director — Cogent Biosciences, Inc.
Locations (6):
- United States (6):
  - Sylvester Comprehensive Cancer Center/ UMHC, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - OSU Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Wagner AJ, Severson PL, Shields AF, Patnaik A, Chugh R, Tinoco G, Wu G, Nespi M, Lin J, Zhang Y, Ewing T, Habets G, Burton EA, Matusow B, Tsai J, Tsang G, Shellooe R, Carias H, Chan K, Rezaei H, Sanftner L, Marimuthu A, Spevak W, Ibrahim PN, Inokuchi K, Alcantar O, Michelson G, Tsiatis AC, Zhang C, Bollag G, Trent JC, Tap WD. Association of Combination of Conformation-Specific KIT Inhibitors With Clinical Benefit in Patients With Refractory Gastrointestinal Stromal Tumors: A Phase 1b/2a Nonrandomized Clinical Trial. JAMA Oncol. 2021 Sep 1;7(9):1343-1350. doi: 10.1001/jamaoncol.2021.2086. PMID 34236401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included a dose escalation portion (Part 1) in which the safety profile and recommended phase 2 dose (RP2D) of CGT9486 as a single oral agent was evaluated in participants with solid tumors (including gastrointestinal stromal tumor [GIST]), followed by signal-seeking extension cohorts of CGT9486 in combination with pexidartinib or sunitinib (Part 2). Parts 2a, 2c, 2d, and 2f were not conducted due to business decisions.
Pre-assignment Details: A total of 51 participants were enrolled; 24 participants were enrolled across 5 cohorts in Part 1, 12 participants were enrolled across 2 cohorts in Part 2b, and 18 participants (including 3 "re-enrolled") were enrolled across 3 cohorts in Part 2e. 1 participant enrolled in Part 1 and 2 participants enrolled in Part 2b and subsequently were re-enrolled in Part 2e with new identification numbers unique to Part 2e. Participant numbers were not reassigned or reused.
Groups:
- Part 1: CGT9486 250 mg QD: Participants received CGT9486 250 milligrams (mg) orally once daily (QD) in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 1: CGT9486 350 mg QD: Participants received CGT9486 350 mg orally QD in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 1: CGT9486 500 mg QD: Participants received CGT9486 500 mg orally QD in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 1: CGT9486 1000 mg QD: Participants received CGT9486 1000 mg orally QD in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 1: CGT9486 500 mg BID: Participants received CGT9486 500 mg orally twice daily (BID) in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting): Participants in fasting condition received CGT9486 500 mg orally QD in combination with pexidartinib 600 mg (administered as 1 capsule of 200 mg in the morning and 2 capsules of 200 mg in the evening) orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting): Participants in non-fasting condition received CGT9486 500 mg orally QD in combination with pexidartinib 600 mg (administered as 1 capsule of 200 mg in the morning and 2 capsules of 200 mg in the evening) orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg: Participants received CGT9486 500 mg orally QD in combination with sunitinib 25 mg orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg: Participants received CGT9486 1000 mg orally QD in combination with sunitinib 25 mg orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg: Participants received CGT9486 1000 mg orally QD in combination with sunitinib 37.5 mg orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
Period: Dose Escalation (up to 670 Days)
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Started | 3 | 4 | 3 | 7 | 7 (1 participant enrolled in Part 1 and subsequently re-enrolled in Part 2e.) | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 3 | 4 | 3 | 7 | 7 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 7 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 3 | 5 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease (Per RECIST) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Dose Extension Part 2b (up to 868 Days)
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Started | 0 | 0 | 0 | 0 | 0 | 4 (2 participants enrolled in Part 2b and subsequently re-enrolled in Part 2e.) | 8 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Progressive Disease (Per RECIST) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Other than specified | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Dose Extension Part 2e (up to 868 Days)
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 10 (2 participants enrolled in Part 2b and 1 participant enrolled in Part 1 and subsequently re-enrolled in Part 2e.)
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 10
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Not completed — Progressive Disease (Per RECIST) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other than specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all participants treated with at least 1 dose of any study drug. Per planned analysis, baseline characteristics data were collected and reported per study part (not per dose group).
Groups:
- Part 1: CGT9486 (Single-Agent): Participants received doses of CGT9486 ranging from 250 to 1000 mg/day orally in 5 sequential dose escalation cohorts (CGT9486 250 mg QD, 350 mg QD, 500 mg QD, 1000 mg QD, and 500 mg BID). Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg: Participants received CGT9486 500 mg orally QD in combination with pexidartinib 600 mg (administered as 1 capsule of 200 mg in the morning and 2 capsules of 200 mg in the evening) orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 2e: CGT9486 + Sunitinib: Participants received CGT9486 500 mg orally QD in combination with sunitinib 25 mg orally, CGT9486 1000 mg orally QD in combination with sunitinib 25 mg orally, or CGT9486 1000 mg orally QD in combination with sunitinib 37.5 mg orally; in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Total: Total of all reporting groups
Arm/Group | Part 1: CGT9486 (Single-Agent) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg | Part 2e: CGT9486 + Sunitinib | Total
Number analyzed (Participants) | 24 | 12 | 15 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.91) | 64.4 (10.43) | 60.1 (9.41) | 60.1 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 8 | 20
  Male | 15 | 9 | 7 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 23 | 11 | 14 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 5
  White | 21 | 9 | 12 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Recommended Phase 2 Dose (RP2D) of CGT9486
Description: RP2D was determined by incidence of dose limiting toxicity (DLT) using Common Terminology Criteria for Adverse Events (CTCAE) V4.03. DLTs: AEs that occurred during Cycle 1, possibly/probably related to study drug, and met 1 of the following criteria: Hematologic Toxicities: Grade 4 neutropenia for >7 days, Grade ≥3 neutropenia with fever, Grade 4 thrombocytopenia, Grade ≥3 thrombocytopenia for >7 days, Grade 4 anemia; Other Toxicities: Any Grade ≥3 (AE or laboratory) toxicity despite adequate supportive care except for following: Grade ≥3 nausea, vomiting, or diarrhea that resolved to Grade ≤2 within 72 hours; Grade 3 fatigue that resolved to Grade ≤2 within 14 days; Grade ≥3 asymptomatic changes in alkaline phosphatase, hypomagnesemia, hyperglycemia, or hypophosphatemia; Grade 3 increases in transaminases for ≤5 days; Any other Grade ≥3 toxicity for which further dose escalation deemed inappropriate.
Time Frame: Cycle 1 of Part 1 (Cycle length = 28 days)
Population: Safety population included all participants treated with at least 1 dose of any study drug.
Measure: Number; unit: mg
Arm/Group | Part 1: CGT9486 (Single-Agent)
Number analyzed (Participants) | 24
mg | 1000

2. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered study drug, which did not necessarily have a causal relationship with the treatment. An AE could be any unfavorable and unintended sign (for example, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not it was considered to be study drug related. This included any newly occurring event or previous condition that had increased in severity or frequency since the administration of study drug. A treatment-emergent AE (TEAE) was an AE that started or worsened in severity on or after the date of the initial dose of study drug. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From the date of first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 670 days)
Population: Safety population included all participants treated with at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: CGT9486 250 mg QD: Participants received CGT9486 250 mg orally QD in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
- Part 1: CGT9486 500 mg BID: Participants received CGT9486 500 mg orally BID in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 7
Participants | 3 | 4 | 3 | 7 | 7

3. Primary Outcome: Part 1: Area Under The Concentration Time Curve From Time Zero to 24 Hours After Dosing (AUC0-24) of CGT9486
Description: AUC0-24 was determined by the linear trapezoidal rule for the ascending portion and by the log trapezoidal rule for the descending portion of the plasma profile. For BID dosing, Cycle 1 Day 15 AUC0-24 was calculated as 2 x area under the concentration time curve from time zero to 12 hours after dosing (AUC0-12). Missing concentration data were excluded from Pharmacokinetic (PK) analysis.
Time Frame: Predose, 1, 3, 5, 7, 9, and 24 hours postdose at Cycle 1 Day 1 and Cycle 1 Day 15
Population: PK population included all participants who had adequate PK data. Here, 'number analyzed signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)*hour/milliliter (mL)
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 7
nanograms (ng)*hour/milliliter (mL)
  Cycle 1, Day 1: number analyzed (Participants) | 3 | 4 | 2 | 7 | 7
  Cycle 1, Day 1 | 9240 (8.7) | 7200 (20.7) | 5980 (41.7) | 11000 (26.3) | NA (NA) — AUC(0-24) on Cycle 1 Day 1 cannot be determined from the 500 mg BID group due to BID dosing (2nd dose given 12 hours after the 1st dose) and limitation of sampling schedule (sampling up to 9 hours after the 1st dose and no samples collected after the 2nd dose).
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 4 | 3 | 6 | 7
  Cycle 1, Day 15 | 18500 (43.7) | 21300 (27.7) | 15400 (65.8) | 22100 (56) | 24800 (51.4)

4. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of CGT9486
Description: Cmax was taken directly from bioanalytical data.
Time Frame: Predose, 1, 3, 5, 7, 9, and 24 hours postdose at Cycle 1 Day 1 and Cycle 1 Day 15
Population: PK population included all participants who had adequate PK data. Here, 'number analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 7
ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 3 | 4 | 2 | 7 | 7
  Cycle 1, Day 1 | 499 (6.92) | 332 (17.9) | 382 (6.48) | 558 (28.1) | 331 (22.8)
  Cycle 1, Day 15 | 869 (38.4) | 1010 (27.5) | 714 (64.9) | 1060 (59) | 1150 (52.4)

5. Primary Outcome: Part 1: Time to Reach Cmax (Tmax) of CGT9486
Description: Tmax was taken directly from merged clinical and bioanalytical data, with time presented as nominal time relative to dose.
Time Frame: Predose, 1, 3, 5, 7, 9, and 24 hours postdose at Cycle 1 Day 1 (Day -10 for 350 mg QD cohort) and Cycle 1 Day 15
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Groups:
- Part 1:CGT9486 500 mg BID: Participants received CGT9486 500 mg orally BID in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1:CGT9486 500 mg BID
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 7
hours
  Cycle 1, Day 1 (or Day -10): number analyzed (Participants) | 3 | 4 | 2 | 7 | 7
  Cycle 1, Day 1 (or Day -10) | 9 [9 to 24] | 16.5 [9 to 24] | 15 [6 to 24] | 9 [3 to 24] | 7 [3 to 9]
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 4 | 3 | 6 | 7
  Cycle 1, Day 15 | 3 [1 to 24] | 9 [0 to 9] | 7 [7 to 24] | 6 [3 to 24] | 5 [1 to 9]

6. Primary Outcome: Part 1: Half Life (T1/2) of PLX9486
Description: Participants in a selected Part 1 cohort (350 mg QD) participated in a PK substudy to obtain more complete information on the PK profile of PLX9486. Participants received a single dose of 350 mg of PLX9486 10 days prior to the start of repeated QD dosing and plasma concentrations were followed 0.5, 1, 2, 4, 6, and 9 hours postdose, and then once daily for 9 additional days prior to Cycle 1 Day 1.
Time Frame: Predose, 0.5, 1, 2, 4, 9, 24, 49, 72, 96, 120, 144, 168, 192, 216 hours postdose on Day -10
Population: Half life of PLX9486 can only be determined in participants who participated in the PK substudy. Sampling schedule in other Part 1 and Part 2 cohorts do not allow for determination of t1/2.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Part 1: CGT9486 350 mg: Participants received a single dose of 350 mg of PLX9486 10 days (on Day -10) prior to the start of 350 mg orally QD in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
Arm/Group | Part 1: CGT9486 350 mg
Number analyzed (Participants) | 4
hours | 75.4 (26.1)

7. Primary Outcome: Part 2e: RP2D of CGT9486 in Combination With Sunitinib
Description: RP2D was determined by incidence of DLT using CTCAE version 4.03 for severity grade. DLTs were defined as AEs that occurred during Cycle 1, classified as possibly/probably related to study drug, and met 1 of the following criteria: Hematologic Toxicities: Grade 4 neutropenia for >7 days, Grade ≥3 neutropenia with fever, Grade 4 thrombocytopenia, Grade ≥3 thrombocytopenia for >7 days or with bleeding, Grade 4 anemia; Other Toxicities: Any Grade ≥3 (AE or laboratory) toxicity despite adequate supportive care except for the following: Grade ≥3 nausea, vomiting, or diarrhea that resolved to Grade ≤2 within 72 hours; Grade 3 fatigue that resolved to Grade ≤2 within 14 days; Grade ≥3 asymptomatic changes in alkaline phosphatase, hypomagnesemia, hyperglycemia, or hypophosphatemia; Grade 3 increases in transaminases for ≤5 days; Any other Grade ≥3 toxicity for which further dose escalation deemed inappropriate.
Time Frame: Cycle 1 of Part 2e (Cycle length = 28 days)
Population: Safety population included all participants treated with at least 1 dose of any study drug.
Measure: Number; unit: mg
Arm/Group | Part 2e: CGT9486 + Sunitinib
Number analyzed (Participants) | 18
mg | 1000

8. Primary Outcome: Part 2b: RP2D of PLX9486 in Combination With Pexidartinib
Description: as for outcome 7
Time Frame: Cycle 1 of Part 2 b (Cycle length = 28 days)
Population: Safety population included all participants treated with at least 1 dose of any study drug.
Measure: Number; unit: mg
Groups:
- Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting): Participants in fasting condition received CGT9486 500 mg orally QD in combination with CGT9486 600 mg (administered as 1 capsule of 200 mg in the morning and 2 capsules of 200 mg in the evening) orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting)
Number analyzed (Participants) | 4 | 8
mg | NA — NA signifies RP2D was not estimable due to no DLTs were experienced during Part 2b. | NA — NA signifies RP2D was not estimable due to no DLTs were experienced during Part 2b.

9. Primary Outcome: Part 2b: Number of Participants With Any TEAEs and Treatment-Related TEAEs
Description: An AE was any untoward medical occurrence in a participant administered study drug, which did not necessarily have a causal relationship with the treatment. An AE could be any unfavorable and unintended sign (for example, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not it was considered to be study drug related. This included any newly occurring event or previous condition that had increased in severity or frequency since the administration of study drug. A TEAE was an AE that started or worsened in severity on or after the date of the initial dose of study drug. Treatment-related TEAEs included all events reported as "possibly related" or "probably related" to any of study treatment. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From the date of first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 868 days)
Population: Safety population included all participants treated with at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting)
Number analyzed (Participants) | 4 | 8
Participants
  TEAEs | 4 | 8
  Related TEAEs | 4 | 7

10. Primary Outcome: Part 2e: Number of Participants With Any TEAEs and Treatment-Related TEAEs
Description: as for outcome 9
Time Frame: From the date of first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 825 days)
Population: Safety population included all participants treated with at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 3 | 5 | 10
Participants
  TEAEs | 3 | 5 | 10
  Related TEAEs | 3 | 5 | 9

11. Secondary Outcome: Part 1: Overall Response Rate (ORR): Percentage of Participants With Best Overall Response of Complete Response (CR) or Partial Response (PR), as Assessed Using RECIST V1.1
Description: ORR was defined as the percentage of participants who achieved a best overall response of confirmed complete response (CR) or partial response (PR). CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of first dose of study drug until the first appearance of CR or PR (maximum exposure: 670 days)
Population: Efficacy evaluable population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline tumor assessment or discontinue study medication early due to disease progression or death.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 6
percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 14.3 [0.4 to 57.9] | 0 [0.0 to 45.9]

12. Secondary Outcome: Part 1: Progression-Free Survival (PFS), as Assessed Using RECIST V1.1
Description: PFS was defined as the number of days from the first day of treatment (Cycle 1 Day 1) to the date of the first documented disease progression or date of death, whichever occurred first. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). The sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions was also considered progression. Median was calculated using Kaplan-Meier estimate.
Time Frame: From the first date of treatment until the first documented disease progression or date of death (maximum exposure: 670 days)
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 6
days | 54 [28 to 56] | 53 [20 to 53] | 48 [47 to 221] | 144 [38 to 335] | 186 [20 to 669]

13. Secondary Outcome: Part 1: Duration of Response (DOR), as Assessed Using RECIST V1.1
Description: DOR was defined as the number of days from the date of first response (PR or CR confirmed at least 28 days later) to the date of first documented disease progression/relapse or death, whichever occurred first. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (target or non-target) must had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions was also considered progression. Median was calculated using Kaplan-Meier estimate.
Time Frame: From the date of first response (PR or CR) to the date of first documented disease progression/relapse or death, whichever occurred first (maximum exposure: 670 days)
Population: Efficacy evaluable population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline tumor assessment or discontinue study medication early due to disease progression or death. Here, 'Overall number of participants analyzed' signifies participants with best overall response of CR or PR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
days |  |  |  | 224 |

14. Secondary Outcome: Part 2: Overall Response Rate (ORR): Percentage of Participants With Best Overall Response of Complete Response (CR) or Partial Response (PR), as Assessed Using RECIST V1.1
Description: ORR was defined as the percentage of participants who achieved a best overall response of confirmed CR or PR. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of first dose of study drug until the first appearance of CR or PR (maximum exposure: 868 days)
Population: Efficacy evaluable population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline tumor assessment or discontinue study medication early due to disease progression or death. Data for 3 re-enrolled participants is included in their initial cohort analysis but not in the Part 2e analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 3 | 8 | 3 | 5 | 7
percentage of participants | 33.3 [0.8 to 90.6] | 0 [0.0 to 36.9] | 33.3 [0.8 to 90.6] | 0 [0.0 to 52.2] | 28.6 [3.7 to 71.0]

15. Secondary Outcome: Part 2: Clinical Benefit Rate (CBR): Percentage of Participants With Clinical Benefit, as Assessed Using RECIST V1.1
Description: Participants were considered to experience clinical benefit if they had a best overall response of stable disease (SD) that lasted for at least 16 weeks, or confirmed best overall response of PR or CR. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters. CR: Disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (target or non-target) must had reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: From the date of first dose of study drug until the first appearance of CR, PR, or SD (maximum exposure: 868 days)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 3 | 8 | 3 | 5 | 7
percentage of participants | 100 [29.2 to 100] | 37.5 [8.5 to 75.5] | 100 [29.2 to 100] | 60.0 [14.7 to 94.7] | 85.7 [42.1 to 99.6]

16. Secondary Outcome: Part 2: Progression-Free Survival (PFS), as Assessed Using RECIST V1.1
Description: as for outcome 12
Time Frame: From the first date of treatment until the first documented disease progression or date of death (maximum exposure: 868 days)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 3 | 8 | 3 | 5 | 7
days | 333 [234 to 336] | 128 [26 to 867] | NA [503 to NA] — Due to smaller number of participants with an event, Median and upper limit of 95% confidence interval (CI) could not be calculated. | 319 [26 to 530] | NA [41 to NA] — Due to smaller number of participants with an event, Median and upper limit of 95% CI could not be calculated.

17. Secondary Outcome: Part 2: Overall Survival
Description: Overall Survival was defined as the number of days from the first day of treatment (Cycle 1 Day 1) until the date of death. If a participant was lost to follow-up, overall survival was censored at the date of last contact. Median was calculated using Kaplan-Meier estimate.
Time Frame: From the first day of treatment until the date of death (maximum exposure: 868 days)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Part 2e:CGT9486 1000 mg QD + Sunitinib 37.5 mg: Participants received CGT9486 1000 mg orally QD in combination with sunitinib 37.5 mg orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e:CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 3 | 8 | 3 | 5 | 7
days | 853 [240 to 853] | 414 [106 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated. | NA [551 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated. | 362 [164 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated. | NA [98 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated.

18. Secondary Outcome: Part 2: Overall Survival at Month 12
Description: Percentage of participants who survived at Month 12 have been reported.
Time Frame: Month 12
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg: Participants received CGT9486 1000 mg QD in combination with sunitinib 37.5 mg orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 3 | 8 | 3 | 5 | 7
percentage of participants | 66.7 [5.4 to 94.5] | 55.6 [7.3 to 87.6] | 100 [100 to 100] | 40.0 [5.2 to 75.3] | 68.6 [21.3 to 91.2]

19. Secondary Outcome: Part 2: PFS at Month 6
Description: PFS was defined as the number of days from the first day of treatment (Cycle 1 Day 1) to the date of the first documented disease progression or date of death, whichever occurred first. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). The sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions was also considered progression. Percentage of participants with PFS at Month 6 are reported.
Time Frame: Month 6
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting): Participants in fasting condition received CGT9486 500 mg QD in combination with pexidartinib 600 mg (administered as 1 capsule of 200 mg in the morning and 2 capsules of 200 mg in the evening) orally in 28-day dosing cycles. Treatment was continued until participant discontinuation, withdrawal, or study termination.
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 3 | 8 | 3 | 5 | 7
percentage of participants | 100 [100 to 100] | 25.0 [1.4 to 63.5] | 100 [100 to 100] | 60.0 [12.6 to 88.2] | 85.7 [33.4 to 97.9]

20. Secondary Outcome: Part 2: Duration of Response (DOR), as Assessed Using RECIST V1.1
Description: as for outcome 13
Time Frame: From the date of first response (PR or CR) to the date of first documented disease progression/relapse or death, whichever occurred first (maximum exposure: 868 days)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 2
days | 169 |  | NA [NA to NA] — Due to smaller number of participants with an event, data could not be calculated. |  | NA [NA to NA] — Due to smaller number of participants with an event, data could not be calculated.

21. Secondary Outcome: Part 2: AUC0-24 of CGT9486 in Combination With Pexidartinib or Sunitinib
Description: AUC0-24 was determined by the linear trapezoidal rule for the ascending portion and by the log trapezoidal rule for the descending portion of the plasma profile. Missing concentration data were excluded from PK analysis.
Time Frame: Predose, 1, 3, 5, 7, 9, and 24 hours postdose at Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 4 | 8 | 3 | 5 | 10
ng*hour/mL
  Cycle 1, Day 1 | 7810 (31.6) | 7910 (21.9) | 9800 (69.4) | 14800 (16.3) | 12700 (28.5)
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 8 | 3 | 5 | 9
  Cycle 1, Day 15 | 20300 (53.2) | 19100 (32.5) | 26500 (61.3) | 41400 (28.9) | 38300 (43.3)

22. Secondary Outcome: Part 2: Cmax of CGT9486 in Combination With Pexidartinib or Sunitinib
Description: Cmax was taken directly from bioanalytical data.
Time Frame: Predose, 1, 3, 5, 7, 9, and 24 hours postdose at Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 4 | 8 | 3 | 5 | 10
ng/mL
  Cycle 1, Day 1 | 384 (34.4) | 412 (26.8) | 512 (69.2) | 866 (10.9) | 681 (28.1)
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 8 | 3 | 5 | 9
  Cycle 1, Day 15 | 991 (53.9) | 924 (30.7) | 1200 (61) | 2040 (13.7) | 1850 (42.5)

23. Secondary Outcome: Part 2: Tmax of CGT9486 in Combination With Pexidartinib or Sunitinib
Description: as for outcome 5
Time Frame: Predose, 1, 3, 5, 7, 9, and 24 hours postdose at Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
Number analyzed (Participants) | 4 | 8 | 3 | 5 | 10
hours
  Cycle 1, Day 1 | 8 [3 to 24] | 9 [5 to 24] | 9 [7 to 9] | 24 [7 to 24] | 9 [7 to 24]
  Cycle 2, Day 15: number analyzed (Participants) | 3 | 8 | 3 | 5 | 9
  Cycle 2, Day 15 | 5 [5 to 9] | 6 [3 to 9] | 3 [0 to 9] | 9 [3 to 24] | 3 [0 to 24]

ADVERSE EVENTS:
Time Frame: From the date of first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 670 days for Part 1; 868 days for Part 2b; 825 days for Part 2e)
Description: Safety population included all participants treated with at least 1 dose of any study drug. One participant enrolled in Part 1 and 2 participants enrolled in Part 2b completed their initial enrollment and subsequently re-enrolled in Part 2e.
Arm/Group | Part 1: CGT9486 250 mg QD | Part 1: CGT9486 350 mg QD | Part 1: CGT9486 500 mg QD | Part 1: CGT9486 1000 mg QD | Part 1: CGT9486 500 mg BID | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/4 | 3/3 | 5/7 | 4/7 | 2/4 | 0/8 | 1/3 | 1/5 | 4/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/4 | 1/3 | 1/7 | 3/7 | 2/4 | 0/8 | 1/3 | 1/5 | 4/10
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 7/7 | 7/7 | 4/4 | 8/8 | 3/3 | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: CGT9486 250 mg QD (N=3) | Part 1: CGT9486 350 mg QD (N=4) | Part 1: CGT9486 500 mg QD (N=3) | Part 1: CGT9486 1000 mg QD (N=7) | Part 1: CGT9486 500 mg BID (N=7) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) (N=4) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) (N=8) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg (N=3) | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg (N=5) | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg (N=10)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prophylaxis against dehydration (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Part 1: CGT9486 250 mg QD (N=3) | Part 1: CGT9486 350 mg QD (N=4) | Part 1: CGT9486 500 mg QD (N=3) | Part 1: CGT9486 1000 mg QD (N=7) | Part 1: CGT9486 500 mg BID (N=7) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Fasting) (N=4) | Part 2b: CGT9486 500 mg QD + Pexidartinib 600 mg (Non-Fasting) (N=8) | Part 2e: CGT9486 500 mg QD + Sunitinib 25 mg (N=3) | Part 2e: CGT9486 1000 mg QD + Sunitinib 25 mg (N=5) | Part 2e: CGT9486 1000 mg QD + Sunitinib 37.5 mg (N=10)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 4 | 1 | 3 | 3 | 2 | 8
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 1 | 0 | 3 | 3 | 2 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 2 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2 | 3 | 4 | 1 | 4 | 2 | 1 | 7
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 3 | 3 | 1 | 2 | 2 | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 2 | 2 | 3 | 1 | 1 | 1 | 1 | 5
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 4 | 2 | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 4
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 4
Weight increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Platelet count increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 3 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 4 | 0 | 4 | 4 | 1 | 4 | 1 | 2 | 4
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 3 | 0 | 3 | 0 | 1 | 2
Pain (General disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Swelling face (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 4 | 1 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3 | 1 | 2 | 2 | 2 | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 0 | 3 | 4
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelash discolouration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0/1 | 0 | 0/2 | 0/0 | 0/1 | 1/2 | 0 | 0/2 | 0/4 — This is a gender specific AE that affects only female participants.
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0/0 | 0/3 | 0/0 | 0/5 | 0 | 0/3 | 1/6 | 0/0 | 0/3 | 0/6 — This is a gender specific AE that affects only male participants.
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0/1 | 0 | 0/2 | 0/0 | 0/1 | 0/2 | 0 | 0/2 | 1/4 — This is a gender specific AE that affects only female participants.
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT02401815/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT02401815/SAP_001.pdf